CLINICAL TRIAL: NCT03831139
Title: What Makes Prevention Work? Cultural Adaptation of an Effective Program for African-American Adolescents
Brief Title: Cultural Adaptation of the TIM&SARA Prevention Program
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID epidemic & measures to control it
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Patrick Possel, Professor, University of Louisville
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 15.0318
Record Dates: First submitted 2019-01-31; First posted 2019-02-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Depressive Symptoms
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prevention (Experimental): TIM&SARA has a duration of 16 fifty-minute sessions and is organized in five modules. The first module (2 sessions) outlines the rationale for the program and establishes connections between group leaders and adolescents. The next module (2 sessions) focuses on helping adolescents to consider already existing goals, set new ones, and learn how to achieve goals to build up the motivation of the youth to learn and apply the material of the following modules. The third module (6 sessions) focuses on understanding the relations among cognitions, emotions, and behaviors, and teaching the participating youths how to identify and challenge negative cognitions. The forth module (5 sessions) trains the youth in assertive and social competent social behavior. Finally, the last session is a review session and includes a celebration. All parts of the program use illustrative, culturally relevant situations introduced by the participating adolescents.
  Interventions: Behavioral: TIM&SARA
- Control (No Intervention): The youth participate in school as usual.

INTERVENTIONS:
Behavioral: TIM&SARA
  Arms: Prevention

SUMMARY:
Disparities between African-American and European-American youth regarding academic outcomes, mental health, and physical health exist. Depression, a very common mental health problem, plays a central role by impacting academic outcomes and cardiovascular health. Thus, a program that successfully reduces the likelihood for youths to develop depression should also reduce problems with academic outcomes and physical health and therefore reduce disparity in all three domains. Research demonstrates that European-American youth benefit more from programs preventing the development of depression than their African-American peers. Thus, the goals of this project are to (a) identify mechanisms that may result in differential program effectiveness across racial groups, and (b) adapt such a program (TIM&SARA) so youth from diverse racial backgrounds benefit similarly. Freshmen in an urban high-school will participate in TIM&SARA, fill out surveys and give biological data in saliva.

DETAILED DESCRIPTION:
Already in adolescence, substantial disparities between African-Americans and European-Americans regarding academic outcomes, mental health, and physical health like cardiovascular health exist. While these domains are often treated as unrelated, they influence each other in a way that the disparity in one variable increases the likelihood for disparity in the others. Depression, a very common mental health problem, plays a central role by impacting academic outcomes and cardiovascular health. Thus, a program that successfully reduces the likelihood for youths to develop depression should also reduce problems with academic outcomes and physical health and therefore reduce disparity in all three domains. Unfortunately, research demonstrates that European-American youth benefit more from programs preventing the development of depression than their African-American peers. Thus, the main goals of this research project are to (a) identify mechanisms that may result in differential prevention program effectiveness across youth race groups, and (b) adapt such a program (TIM&SARA) so youth from diverse racial backgrounds benefit similarly.

In this project, the depression prevention program TIM&SARA will be implemented as part of the normal school curriculum for freshmen in an urban high-school. The differential effects of the program on African-American and European-American youths will be examined using surveys and biological data in saliva.

ELIGIBILITY:
Inclusion Criteria:

* 9th grade students in the participating high school

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 740 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Center for Epidemiological Studies - Depression Scale (CES-D) | 5 minutes
  The CES-D is a 20-item self-report instrument which has been repeatedly used in adolescent samples (e.g., Roberts et al., 1990) will be used. Items are rated on a 4-point Likert scale (0 = rarely or none of the time; 3 = most of the time; e.g., "I was bothered by things that usually don't bother me."). The scale ranges from 0-60; total scores of 16 or higher indicate clinically significant depressive symptoms. The internal consistency of the CES-D in previous studies with adolescents is good (α = .92, Winkeljohn Black, & Pössel, 2015).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Possel, Dr.rer.soc., Principal Investigator — University of Louisville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seely HD, Possel P. Equity and inclusion in prevention: Depression prevention in Black and White American youth. J Consult Clin Psychol. 2025 Apr;93(4):307-316. doi: 10.1037/ccp0000918. PMID 40126558